CLINICAL TRIAL: NCT00177827
Title: Voriconazole Prophylaxis Against Aspergillosis in Lung Transplant Recipients: Pharmacokinetics and Correlation Between Plasma and Lung Concentrations With Toxicity/Efficacy
Brief Title: Voriconazole Prophylaxis Against Aspergillosis in Lung Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: IRB# 0304017
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2009-12-03 (Estimated); Status verified 2009-12

CONDITIONS: Post Lung Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A fixed dosage regimen of voriconazole is routinely used for prophylaxis of aspergillosis in lung transplant patients at our institution. We hypothesize that use of a fixed dosage voriconazole regimen leads to large degree of variability in drug exposure among lung transplant patients and consequently, therapeutic failures or toxicity. This is a three part study which will examine plasma and lung voriconazole concentrations achieved with the prophylactic regimen and assess for a correlation between these concentrations with efficacy and toxicity. We aim to conduct an initial pilot study in 12 lung transplant patients to characterize the pharmacokinetic profile of voriconazole with both intravenous and oral doses. The data gathered from the pilot pharmacokinetic study will then be utilized to correlate trough concentrations with total voriconazole drug exposure as measured by area under the plasma concentration versus time curve (AUC). Additionally, trough concentrations will be followed over nine weeks of the prophylactic treatment period in a larger cohort of patients to determine maintenance of consistency in trough concentrations and whether the plasma concentrations are predictive of efficacy and toxicity. Voriconazole lung concentrations will be measured in a pilot study of 12 patients who undergo a bronchoscopy procedure as part of their standard medical care in order to determine the relationship between plasma and lung concentrations. The information obtained from this three phase study will be utilized to characterize the pharmacokinetics of voriconazole in lung transplant patients. Further, it will be used to define an optimal therapeutic voriconazole regimen that will be individualized to target specific concentrations in the lung and plasma to maximize efficacy and minimize toxicity

DETAILED DESCRIPTION:
Blood samples (5 mL) will be collected either from an existing indwelling intravenous catheter or via a catheter placed by a research nurse or phlebotomist. The samples will be centrifuged at 1,500 g for 10 minutes within 60 minutes of collection. The plasma will be separated into two separate cryovials and stored at - 80 C until the time of assay for Voriconazole.A standardized data collection sheet will be created by the study investigators and utilized to gather pertinent information on each study participant from the patient medical records and electronic databases. The type of information collected will include, but will not be limited to, demographic information, transplant history, periodic serum chemistry and hematology monitoring, medication regimen, plasma voriconazole level monitoring and efficacy and safety monitoring parameters.

ELIGIBILITY:
Inclusion Criteria:

* Male or female lung transplant recipients, greater than 18 years old, who are initiated on the voriconazole prophylactic regimen (Figure 1) by their transplant physician as standard care will be eligible for inclusion in the study.

Exclusion Criteria:

* Patients receiving voriconazole to treat an active fungal infection will be excluded. Patients that are concurrently receiving medications that are documented to affect voriconazole pharmacokinetics will be excluded. The agents included, but may not be limited to the following ;carbamazepine, phenytoin, omeprazole, rifabutin and rifampin.10

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chart review
Sampling Method: Probability Sample
Enrollment: 104
Dates: Start 2004-03; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Blair Capitano, Pharm D, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States